CLINICAL TRIAL: NCT02010879
Title: The Impact of Platelet Count, Platelet Mass Index and Platelet Function Evaluated by Platelet Function Analyzer (PFA-100) on Spontaneous Ductal Closure in Preterm Infants
Brief Title: The Impact of Platelet Functions on Spontaneous Ductal Closure in Preterm Infants
Acronym: PFA100
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Omer Erdeve, Associate Professor, Ankara University
Other Study IDs: PDAPFA-100 TRIAL
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Patent Ductus Arterioses
Keywords: patent ductus arterioses; ductal closure; thrombocyte

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although thrombocytopenia has been reported as a risk factor for patent ductus arterioses, there is lack of data on the function of platelets in ductal closure. Information on functions of platelets in ductal closure may change the known model for ductus arterioses and may affect the treatment modalities.

DETAILED DESCRIPTION:
Patent ductus arterioses is a common problem which involves both pulmonary and cardiac outcomes in preterm infants. Although thrombocytopenia has been reported as a risk factor for patent ductus arterioses, there is lack of data on the function of platelets in ductal closure.

The investigators aim to investigate the relation between thrombocytopenia and platelet functions in pathogenesis of spontaneous ductal closure. The investigators hypothesize that Information on functions of platelets in ductal closure may change the known model for ductus arterioses and may affect the treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* gestational age lower than 30 weeks and birth weight lower than 1500 g
* obtained informed consent

Exclusion Criteria:

* any received medical treatment in first 2 days of life
* death in first 2 days
* patients who received any thrombocyte or fresh frozen plasma suspensions
* any known genetic thrombocyte disorder in the family

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: preterm infants with gestational age below 30 weeks and birth weght lower than 1500 g
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
spontaneous ductal closure | 8 weeks
  ductal closure confirmed by echocardiography on postnatal 2-3 days

SECONDARY OUTCOMES:
need for treatment | 8 weeks
  any need for medical treatment (ibuprofen or paracetamol) or surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Omer Erdeve, Professor, Principal Investigator — Ankara University
Locations (1):
- Ankara University Children's Hospital, Ankara, Ankara, Turkey (Türkiye)